CLINICAL TRIAL: NCT00307242
Title: A Single Center Open-Label, Randomized Study Comparing the Safety of Immediately Switching From Lamivudine to Adefovir Dipivoxil Versus Overlapping Lamivudine and Adefovir for 12 Weeks Before Instituting Adefovir Dipivoxil Monotherapy in Patients With Chronic Hepatitis B
Brief Title: Study Comparing the Safety of Switching From Lamivudine to Adefovir Dipivoxil Versus Overlapping Lamivudine and Adefovir Before Adefovir Dipivoxil Monotherapy in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05U.164
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Chronic Hepatitis B
Keywords: Adefovir Dipivoxil; Lamivudine; Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Direct switch to Adefovir Dipivoxil from Lamivudine (Active Comparator)
  Interventions: Drug: Adefovir Dipivoxil
- Overlapping Lamivudine and Adefovir Dipivoxil for 3 months followed by ADV monotherapy (Active Comparator)
  Interventions: Drug: Adefovir Dipivoxil

INTERVENTIONS:
Drug: Adefovir Dipivoxil

SUMMARY:
In earlier clinical studies, when patients who have been on lamivudine (LAM) were switched to adefovir dipivoxil (ADV), some patients developed ALT flares with an elevation of ALT > 10 x the upper limits of normal (ULN).

There were no cases of hepatic decompensation with the flares, however. The transition methods were varied among physicians from no overlapping to overlapping for 1 to 3 months with LAM and ADV. There is still some uncertainty about the optimal approach to switching from LAM to ADV.

This study will compare the safety of directly switching to ADV to a protocolled switch after a period of overlap of 12 weeks. This will facilitate pro-active switching in patients on LAM and will also highlight genotypic resistance ahead of phenotypic resistance as a reason to switch patients. Data to date have only been presented as part of a controlled study in patients with clinically evident LAM-resistance. This study will enroll patients who still have serum hepatitis B virus (HBV) DNA suppression whilst receiving LAM.

DETAILED DESCRIPTION:
Chronic HBV infection is an important worldwide cause of morbidity, mortality and source of potential new infections. There are an estimated 350 million carriers of HBV in the world. In China, Southeast Asia and sub-Saharan Africa, as many as 10-15% of the population are chronically infected. In North America and Northern Europe, infection and carrier rates are much lower, usually below 1%. Intermediate carrier rates of 1-5% are found in Southern Europe (e.g., Italy, Greece and Spain), parts of South and Central America, the Middle East and Japan. Persistent infection develops in over 90% of perinatally infected children and in 3-10% of people who become infected after the age of 6 years. Worldwide, it has been estimated that more than one million people die annually due to HBV-related end stage diseases such as cirrhosis and hepatocellular carcinoma.

The goal of antiviral therapy for hepatitis B is to reduce a patient's risks for progressive liver disease through prolonged suppression or eradication of HBV infection and to arrest or ameliorate HBV-related liver damage.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age with chronic hepatitis B
* Hepatitis B surface antigen (HBsAg)(+) for a minimum of 6 months prior to entry
* Hepatitis B envelope antigen (HBeAg)(+) or (-) at baseline
* Patients having previously received LAM for at least 24 weeks
* Patients with compensated liver function (Child-Pugh score ≤ 6)

Exclusion Criteria:

* Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol.
* Received immunoglobulins, interferon or other immune or cytokine-based therapies with possible activity in hepatitis B disease within 6 months prior to study screening.
* Organ or bone marrow transplant recipients.
* Evidence of active liver disease due to other causes (e.g., Wilson's disease, hemochromatosis, autoimmune hepatitis, hepatitis C or hepatitis D co-infection)
* Patients taking parenteral (intravenous or intramuscular or subcutaneous) or oral steroids, immuno-suppressant therapies or chemotherapeutic agents within 2 months of study screening or expected to receive these agents during the course of the study.
* Previous participation in an investigational trial involving administration of any investigational compound within 2 months prior to the study screening or those who received anti-HBV therapy other than lamivudine within the previous 3 months (e.g. anabolic steroids, ketaconazole, itraconazole, isoniazid, rifampin, rifabutin, simvastatin, lovastatin)
* Clinically relevant alcohol or drug use or history of alcohol or drug use considered by the investigator to be sufficient to hinder compliance with treatment, follow up procedures or evaluation of adverse events
* Lactating females or females with a positive serum pregnancy test.
* Females of childbearing potential (post-puberty) unwilling or unable to have pregnancy testing at any study visit
* Therapy with nephrotoxic drugs (e.g. aminoglycosides, amphotericin B, vancomycin, cidofovir, foscarnet, cisplatin pentamidine, tacrolimus, cyclosporine) or competitors of renal excretion (e.g. probenecid) within 2 months prior to study screening or the expectation that subject will receive these during the course of the study.
* The use of antiviral therapy with agents demonstrating potential anti-HBV activity other than lamivudine within the previous 3 months (e.g. famciclovir, lobucavir, emtricitabine, DAPD, L-FMAU, entecavir, ganciclovir or others).
* History of hypersensitivity to nucleoside and/or nucleotide analogues.
* Clinical, ultrasonographic or radiologic evidence of hepatic mass suggestive of hepatocellular carcinoma.
* Serum alphafetoprotein (AFP) > 50 ng/mL at the first screening visit. However, if the AFP level is > 50 ng/mL at the first screening visit, but has remained stable or decreased over the 6 months preceding the first screening visit, and if there is no radiologic or ultrasonic evidence of hepatic mass(es) suggestive of hepatocellular carcinoma, the patient will be allowed to enroll.
* Inability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06-17 (Actual); Primary Completion 2009-02 (Actual); Study Completion 2009-02-05 (Actual)

PRIMARY OUTCOMES:
Observe the proportion of patients with ALT elevations (> 10 x ULN) at any time over the course of the switch | baseline, 3, 6, 9, and 12 months
Study serum HBV DNA levels over time | baseline, 3, 6, 9, and 12 months
Study serum ALT levels over time | baseline, 3, 6, 9, and 12 months
Study the proportion of patients with YMDD variants at entry | baseline, 3, 6, 9, and 12 months
Study the safety during the switching period | baseline, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hie-Won Hann, M.D., Principal Investigator — Thomas Jefferson University